CLINICAL TRIAL: NCT06566833
Title: Effectiveness of Different Remineralizing Strategies on the Management of Early Carious Lesions in Primary Teeth (Randomized Controlled Clinical Trial)
Brief Title: Effectiveness of Different Remineralizing Strategies on the Management of Early Carious Lesions in Primary Teeth
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Sarah Khairy, assistant lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00010556 - IORG 0008839
Record Dates: First submitted 2024-08-09; First posted 2024-08-22 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: White Spot Lesion
Keywords: curodont repair fluoride plus; CPP-ACPF; sodium fluoride varnish; guided enamel regeneration
MeSH Terms: interventions — Fluorides; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- curodont repair fluoride plus (Experimental): self-assembling peptide (p11-4) with 0.05% sodium fluoride
  Interventions: Drug: self assmbling peptide p11-4 combined with 0.05% fluoride
- CPP-ACPF varnish (Experimental): casein phoshphopeptide amorphous calcium phosphate fluoride (CPP-ACPF )
  Interventions: Drug: Casein phosphopeptide amorphous calcium phosphate
- 5 % sodium fluoride varnish (Active Comparator): 5% sodium fluoride varnish
  Interventions: Drug: 5% sodium fluoride varnish

INTERVENTIONS:
Drug: self assmbling peptide p11-4 combined with 0.05% fluoride — biomimetic remineralizing agent
  Other Names: SAP P11-4
  Arms: curodont repair fluoride plus
Drug: Casein phosphopeptide amorphous calcium phosphate — remineralizing agents that acts as a fluoride booster
  Other Names: CPP-ACPF
  Arms: CPP-ACPF varnish
Drug: 5% sodium fluoride varnish — remineralizing agent that is used as a gold standard for remineralization
  Other Names: 5% NaF
  Arms: 5 % sodium fluoride varnish

SUMMARY:
the primary aim of the study is remineralization of early carious lesions in primary teeth using different remineralizing agents of different remineralizing strategies when applied in an intensive mode. The secondary aim of the study is to compare their antibacterial effect against streptococcus mutans and their effect on reducing the size of the lesions.

DETAILED DESCRIPTION:
The primary aim of the study is to compare the effect of curodont repair fluoride plus (self-assembling peptide p11-4 with 0.5% sodium fluoride) with MI varnish (casein phosphopeptide amorphous calcium phosphate fluoride) and Colgate fluoride varnish (5% sodium fluoride) in remineralization of early carious lesions in primary anterior teeth. The study sample is consisted of 66 patients aged 3-6 years old with at least 2 white spot lesions in their primary anterior teeth who are assigned into control group (n=22): colgate fluoride varnish, test group 1(n=22): MI varnish and test group 2 (n=22) :curodont repair fluoride plus. Each material is applied once every 2 weeks for 3 times (intensive mode of application). The secondary aim of the study is to determine the antibacterial effect of each material against streptococcus mutans is compared by obtaining a plaque sample at baseline then after application by 48 hours, 1 months and 3 months and culturing using disk diffusion method for determining the log count of streptococcus mutans at each time point. Another secondary aim is to determine the change in lesion size at baseline and after 6 months and 12 months using standardized photographs with a digital camera.

ELIGIBILITY:
Inclusion Criteria:

1. healthy children
2. age range 3-6
3. at least 2 early carious lesions

Exclusion Criteria:

1. Children presenting with special health care needs or undergoing medical treatment for chronic or acute diseases.
2. Application of fluoride varnish less than 3 months prior to study treatment.
3. Any metabolic disorders affecting bone turnover.
4. Concurrent participation in another clinical trial.
5. Patients receiving any antibiotic within 1 month prior to plaque sample collection

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Assessing the remineralization of early carious lesions in primary teeth | 3,6,9 and12 months
  comparing the remineralization effect of different remineralizing agents both qualitatively by comparing the change in ICDAS -11 criteria and quantitatively by using laser fluorescence scores using kavo DIAGNOdent classic after intensive mode of application of the different remineralizing agents

SECONDARY OUTCOMES:
comparing the change in esthetic appearance of early carious lesion before and after treatment | 12 months
  comparing the change in lesion size using standardized photographs quantitatively by calculating pixel size of the lesion before treatment and after 6 and 12 months of intensive mode of application of the different remineralizing agents using ImageJ software program for image analysis. Assessing the esthetic appearance of the lesions will be done subjectively by using a visual analogue scale score from 1 to 7
comparing the antibacterial effect of different remineralizing agents against streptococcus mutans | 3 months
  Supragingival plaque samples will be collected at baseline then after 48 hours, 1 months and 3 months of application of the materials in an intensive mode. log count of streptococcus mutans is determined using disk diffusion method using mitis salivaris agar plates

CONTACTS AND LOCATIONS:
Overall Officials: karin dowidar, professor, Study Director — faculty of Dentistry, Alexandria university, Egypt
Locations (1):
- Karin Dowidar, Alexandria, Professor, Egypt

IPD SHARING:
Plan to Share IPD: No
only the results of the primary and secondary outcomes of the study will be published after study completion

REFERENCES:
- [Background] Mekky AI, Dowidar KML, Talaat DM. Casein Phosphopeptide Amorphous Calcium Phosphate Fluoride Varnish in Remineralization of Early Carious Lesions in Primary Dentition: Randomized Clinical Trial. Pediatr Dent. 2021 Jan 15;43(1):17-23. PMID 33662244